CLINICAL TRIAL: NCT00001615
Title: Phase I Study of Corticosteroid Treatment of Ill-Defined Choroidal Neovascularization in Age-Related Macular Degeneration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 970151; 97-EI-0151
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-05

CONDITIONS: Choroidal Neovascularization; Macular Degeneration
Keywords: Age-Related Macular Degeneration; Choroidal Neovascularization; Disciform; Drusen; Natural History; Periocular; Quality of Life; Steroids; Corticosteroid
MeSH Terms: conditions — Choroidal Neovascularization; Macular Degeneration | interventions — Adrenal Cortex Hormones

INTERVENTIONS:
Drug: Corticosteroid

SUMMARY:
Age-related macular degeneration (AMD) represents the most common cause of blindness in patients over the age of 60. The major cause of vision loss in this disease is due to the development of choroidal neovascular membrane formation (CNVM). Several clinical trials have proven that eyes with "well-defined" CNVM or lesions that can be readily demarcated with fluorescein angiography can be successfully treated with laser photocoagulation. However, up to 87% of eyes present with "ill-defined" CNVM or lesions that cannot be well demarcated on fluorescein angiography and are not amenable to laser photocoagulation. No beneficial treatment for this form of choroidal neovascularization has been established.

Histopathologic study has demonstrated the presence of inflammatory and reparative responses in the retina of patients with ill-defined choroidal neovascularization. Since corticosteroids have been shown to downregulate many of the cellular factors involved in both inflammation and repair, the present study is designed to assess the ability of corticosteroid injection around the eye to prevent severe vision loss associated with "ill-defined" choroidal neovascularization in the setting of age-related macular degeneration. The study will be organized as a randomized open label control clinical trial involving 2 phases. Phase 1 involving 40 patients will establish the feasibility and safety of this treatment modality. Phase 2 will place emphasis on efficacy of the study.

DETAILED DESCRIPTION:
Age-related macular degeneration (AMD) represents the most common cause of blindness in patients over the age of 60. The major cause of vision loss in this disease is due to the development of choroidal neovascular membrane formation (CNVM). Several clinical trials have proven that eyes with "well-defined" CNVM or lesions that can be readily demarcated with fluorescein angiography can be successfully treated with laser photocoagulation. However, up to 87% of eyes present with "ill-defined" CNVM or lesions that cannot be well demarcated on fluorescein angiography and are not amenable to laser photocoagulation. No beneficial treatment for this form of choroidal neovascularization has been established.

Histopathologic study has demonstrated the presence of inflammatory and reparative responses in the retina of patients with ill-defined choroidal neovascularization. Since corticosteroids have been shown to downregulate many of the cellular factors involved in both inflammation and repair, the present study is designed to assess the ability of corticosteroid injection around the eye to prevent severe vision loss associated with "ill-defined" choroidal neovascularization in the setting of age-related macular degeneration. The study will be organized as a randomized open label control clinical trial involving 2 phases. Phase 1 involving 40 patients will establish the feasibility and safety of this treatment modality. Phase 2 will place emphasis on efficacy of the study.

ELIGIBILITY:
Diagnosis of AMD defined by the presence of drusen in one eye and age over 50.

Vision 20/400 or worse in the fellow eye due to exudative complications from CNVM under the fovea.

Visual acuity of 20/80 - 20/200 in the study eye.

Ineligibility for a clinically proven laser photocoagulation protocol.

No patients with age less than 50.

No patients with previous laser therapy for surgery for choroidal neovascularization in the study eye.

No patients with choroidal neovascularization, in the study eye, associated with other ocular diseases such as pathologic myopia, ocular histoplasmosis, posterior uveitis, idiopathic, etc.

No patients with presence of geographic atrophy or serous pigment epithelial detachment under the fovea in the study eye.

No patients with decreased vision, in the study eye, due to retinal disease not attributable to ill-defined CNVM, such as serous retinal pigment epithelial detachment, nonexudative form of ARM, geographic atrophy, inherited retinal dystrophy, uveitis, epiretinal membrane and others.

No patients with decreased vision, in the study eye, due to significant media opacity such as corneal disease or cataract.

No patients with systemic or local therapy that may alter the natural course of ill-defined CNVM, especially antiangiogenic treatment with thalidomide or alpha interferon.

No patients with intraocular pressure greater than or equal to 26 or history suggesting glaucoma (e.g., history of the diagnosis of glaucoma, past or present use of medications to control intraocular pressure, or disc/nerve fiber layer defects suggestive of glaucoma) and glaucomatous visual field defects as documented by Goldmann or Humphrey perimetry taken within 6 months to qualification.

No patients with any contraindications to performing the necessary diagnostic studies, especially the use of fluorescein angiography.

No patients with known history of untoward complications from corticosteroid therapy, including elevated intraocular pressure in response to topical or periocular corticosteroids.

No patients with medical problems which make consistent follow-up over the treatment period unlikely (e.g., stroke, severe MI, terminal carcinoma.

No patients with current use of or likely need for systemic or ocular medications known to be toxic to the lens, retina or optic nerve, such as: Deferoxamine, Chloroquine/Hydroxychloroquine (Plaquenil), Tamoxifen, Chlorpromazine, Phenothiazines, Ethambutol, Ocular or systemic steroids or use of steroid-containing inhalers or nasal sprays utilized more than 6 days a month on average-any regular use of pills containing steroids.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180
Dates: Start 1997-07; Study Completion 2000-05

CONTACTS AND LOCATIONS:
Locations (1):
- National Eye Institute (NEI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Dastgheib K, Green WR. Granulomatous reaction to Bruch's membrane in age-related macular degeneration. Arch Ophthalmol. 1994 Jun;112(6):813-8. doi: 10.1001/archopht.1994.01090180111045. PMID 7516148
- [Background] Bressler NM, Maguire MG, Murphy PL, Alexander J, Margherio R, Schachat AP, Fine SL, Stevens TS, Bressler SB. Macular scatter ('grid') laser treatment of poorly demarcated subfoveal choroidal neovascularization in age-related macular degeneration. Results of a randomized pilot trial. Arch Ophthalmol. 1996 Dec;114(12):1456-64. doi: 10.1001/archopht.1996.01100140654002. PMID 8953976